CLINICAL TRIAL: NCT04736641
Title: Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: 26.01.2021-E.13996
Record Dates: First submitted 2021-01-30; First posted 2021-02-03 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Hip Disease; Hip Pain Chronic
Keywords: Hip disease; Reliability; Validity; Cross-cultural adaptation
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Individuals with hip disease and chronic pain on hip
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire (JOAHDEQ) will be applied

SUMMARY:
The purpose of this study was to investigate adaptation, validity, and reliability of the Turkish version of the Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire (JOAHDEQ).

DETAILED DESCRIPTION:
There are a number of medical assessment tools for various diseases, but in most cases such tools are designed to reflect the perspective of healthcare providers, not perspective of patients. In addition to clinical results, it is necessary to evaluate the quality of life of patients when measuring the effect of medical treatments. Thus, evaluation criteria which can be useful as patient-reported outcome indices, have received increasing attention in recent years. Health-related quality of life provides a patient-reported assessment. Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire (JOAHDEQ) evaluates quality of life related to hip disorders. It is also a guide in determining the expectations of individuals in the treatment process. It consists of 3 subscales (pain, movement and mental) and 20 items. Hip condition and pain are evaluated with a 100 mm scale. 20 items are scaled likert with values between 0 and 4. "0" means "strongly agree", "1" means "agree", "2" means "uncertain", "3" means "disagree" and "4" means "strongly disagree". The study is planned with 105 individuals with hip disease. After questioning the sociodemographic characteristics of the individuals, the patients will be asked to fill in JOAHDEQ, Oxford Hip Score, International Hip Outcome Tool-12, Short Form-36, and Visual Analog Scale Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Any diagnosed hip disease,
* Chronic hip pain,
* History of pain when lying or during weight-bearing activities, aggravated by activity for more than 3 months.

Exclusion Criteria:

* Lumbar spine nerve root findings,
* History of lumbar spine or hip surgery,
* Corticosteroid injection to hip in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with hip disease and chronic pain on hip.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire (JOAHDEQ) | 15 minutes
  Japanese Orthopaedic Association Hip Disease Evaluation Questionnaire is designed to evaluate quality of life related to hip disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR